CLINICAL TRIAL: NCT01310933
Title: Ultrasonographic Differentiation Between Kikuchi's Disease and Lymphoma in Patients With Cervical Lymphadenopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Jen Liao, Department of Otolaryngology, Far Eastern Memorial Hospital
Other Study IDs: 099086-E
Record Dates: First submitted 2011-02-21; First posted 2011-03-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Lymphoma; Kikuchi's Disease
MeSH Terms: conditions — Lymphoma; Histiocytic Necrotizing Lymphadenitis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kikuchi's disease
- Malignant lymphoma

SUMMARY:
The purpose of this study is to differentiate Kikuchi's disease and malignant lymphoma by soft tissue ultrasound.

DETAILED DESCRIPTION:
Introduction Kikuchi's disease (KD) is a histiocytic necrotizing lymphadenitis that was described for the first time in Japan in 1972 almost simultaneously by Kikuchi and Fujimoto1-2. KD is a self-limited necrotizing lymphadenitis and occurs predominantly in females between 20 and 30 years old. Its main presentation is cervical lymphadenopathy. The diagnosis of KD is based on clinical manifestation, fine-needle aspiration cytology or excision biopsy. The pathological characteristics include patchy paracortical lymphohistiocytic aggregates with variable karyorrhexis and absence of granulocytic infiltration. Antibiotics are not helpful symptoms remit within six months spontaneously.

As KD is a benign and self-limiting disease, proper diagnosis may help avoid unnecessary treatment. KD can be easily confused clinically, pathologically, and radiologically with malignant lymphadenopathy, especially lymphoma. Several reports have described the CT characteristics of KD3-4, including enlarged, multiple lymph nodes that are homogeneously enhanced without evidence of gross necrosis. The CT appearance of Kikuchi's disease may be variable, thus mimicking lymphoma4. In previous work, the ultrasound appearance of KD has not been well-described and has been compared to lymphoma. In this study, we compared the sonographic characteristic of Kikuchi's disease and malignant lymphoma.

Patients and methods From November 2007 to September 2009, sonograms of twelve case notes with pathological diagnoses of Kikuchi's disease and twelve patients with malignant lymphoma were studied.

The sonograms were performed by the same sinologist (L-J Liao) using an ATL HDI 5000 with a high-resolution 7.5- to 12-MHz real-time linear-array transducer (Philips Ultrasound, Bothell, WA, USA). Morphological US parameters were thoroughly evaluated and recorded on the Marosis PACS system (Marotech Inc., Seoul, South Korea). The lengths of short and long axes of enlarged lymph nodes were measured and recorded. The shape of the lymph node was determined by the short axis to long axis ratio (S/L ratio). The nodal border was assessed for sharpness. Echogenicity of the lymph nodes was compared with that of adjacent muscles. Swelling of the surrounding tissues that presented with hyperechoic rims was assessed. The nodes were considered matted when a number of lymph nodes were clustered together. The internal architecture of lymph nodes was examined for the presence of heterogeneous micronodular pattern or reticulation.

Fisher's exact test and X 2 test were used to calculate the significance of the difference in gray-scale features. Mann-Whitney U tests were used to calculate the significance of the difference in nodal size and short- to long-axis ratio.

Expected Results:

We suppose that basic ultrasonographic characteristics (size, shape, rims, matting, and micronodular echotexture) help in the differentiation of cervical lymph nodes in patients with Kikuchi's disease and lymphoma. A precise diagnosis of KD is possible avoiding unnecessary biopsies or aggressive treatment.

References:

1. Kikuchi M. Lymphadenitis showing focal reticulum cell hyperplasia with nuclear debris and phagocytosis. Nippon Ketsueki Kakkai Zasshi 1972;35:379-80.
2. Fujimoto Y, Kozima Y, Yamaguchi K. Cervical subacute necrotizing lymphadenitis. A new clinicological entity. Naika 1972;376:247-53.
3. Kwon S, Kim T, Kim Y, Lee K, Lee N, Seol H. CT findings in Kikuchi disease: analysis of 96 cases. American Journal of Neuroradiology 2004;25(6):1099.
4. Na D, Chung T, Byun H, Kim H, Ko Y, Yoon J. Kikuchi disease: CT and MR findings. American Journal of Neuroradiology 1997;18(9):1729.

ELIGIBILITY:
Inclusion Criteria:

From November 2007 to September 20010, pathological diagnoses of Kikuchi's disease & malignant lymphoma were studied sonograms available

Exclusion Criteria:

no pathology no sonograms

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From November 2007 to September 20010, sonograms of eleven cases notes with pathological diagnoses of Kikuchi's disease and ten patients with malignant lymphoma were studied.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Liao, MD, Study Chair — Department of Otolaryngology Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan, Pan Chiao, Taipei, Taiwan